CLINICAL TRIAL: NCT06076746
Title: Evaluation of Psychotherapeutic Intervention Model in Nursing on Patients With Nursing Diagnosis of Ineffective Coping
Brief Title: Evaluation of Psychotherapeutic Intervention Model in Nursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuğba Aşkan (Other)
Responsible Party: Sponsor-Investigator, Tuğba Aşkan, Nurse, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1081
Record Dates: First submitted 2023-05-09; First posted 2023-10-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-10

CONDITIONS: Anxiety Generalized
Keywords: Nursing Outcomes Classification; Psychotherapeutic intervention; Patient outcome; Psychiatric nursing; Anxiety Generalized; Coping; Self esteem
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: It will not be known by the Outcomes Assessor that the patients are in the experimental or usual treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Intervention(s) for ineffective coping in General Anxiety (Experimental): Patients with nurse diagnosis of ineffective coping will be treated using Nursing Interventions Classification (NIC) psychotherapeutic intervention(s).
  Interventions: Behavioral: NIC Psychotherapeutic Intervention(s) for İneffective Coping; Behavioral: psychotherapeutic intervention
- Treatment-as-Usual for General Anxiety (Active Comparator): Patients with nurse diagnosis of ineffective coping will receive the usual treatment for general anxiety.
  Interventions: Behavioral: psychotherapeutic intervention

INTERVENTIONS:
Behavioral: NIC Psychotherapeutic Intervention(s) for İneffective Coping — Patients will be treated by NIC psychotherapeutic intervention(s) for general anxiety (e.g. anxiety reduction, coping enhancement).
  Arms: Experimental: Intervention(s) for ineffective coping in General Anxiety
Behavioral: psychotherapeutic intervention — Patients will be treated by NIC psychotherapeutic intervention(s) for general anxiety (e.g. anxiety reduction, coping enhancement).

SUMMARY:
This study aims to evaluate the efficacy of a psychotherapeutic intervention model in nursing on the nursing diagnosis ineffective coping. For this purpose, validity and reliability studies of the assessment tools will be carried out initially, and then a randomized controlled study will be conducted.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy of the psychotherapeutic intervention model in nursing on patients with nursing diagnosis of ineffective coping (International Classification of Nursing Practices (ICNP)/North American Nursing Diagnostic Association (NANDA)). For this purpose, first of all, validity and reliability studies of "Coping" and "Self-Esteem", which are the results of NOC (Nursing Outcomes Classification), will be conducted, and then a randomized controlled study will be conducted (Turkish version). 200 patients will be included in the validity and reliability phase of the study, which was conducted in a hospital outpatient psychiatric setting in Turkey. The randomized controlled second phase will be carried out, single-blind, nurse-led, with approximately 20 patients with anxiety randomized to intervention (n=10) or control groups (n=10). The usual treatment and care will be compared with the application of the psychotherapeutic intervention model previously developed in nursing.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old,
* Literacy,
* Having applied to the psychiatry outpatient clinic,
* Being regularly treated in a psychiatry outpatient clinic,
* Having a medical diagnosis of generalized anxiety disorder,
* Having at least one of the defining characteristics of the nursing diagnosis of ineffective coping according to the nursing process.

Exclusion Criteria:

* Medical diagnosis of dementia or psychotic spectrum disorder,
* Cognitive disorder,
* Confused state of consciousness
* Psychomotor agitation,
* Moderate or severe intellectual disability
* Expressing suicidal thoughts
* Suicide attempt in the last month
* Continuing psychological counseling at the moment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Coping | Baseline and through study completion, an average of 9 weeks
  Nursing Outcomes Classification (Coping (1302)) The scale consists of 19 items. A minimum of 19 and a maximum of 95 points can be obtained from the scale. Increasing scale scores indicate good results.
Self esteem | Baseline and through study completion, an average of 9 weeks
  Nursing Outcomes Classification (Self-Esteem (1205)) The scale consists of 20 items. A minimum of 20 and a maximum of 100 points can be obtained from the scale. An increase in scale scores indicates good results.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Aşkan, PhD Student, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Çubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided